CLINICAL TRIAL: NCT04944134
Title: Vaccine Ig Levels in Nasal Mucosa as Measured by Nasal Epithelial Lining Fluid
Brief Title: COVID-19 Antibody Levels After Vaccines
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 21-0371
Record Dates: First submitted 2021-06-25; First posted 2021-06-29 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-05

CONDITIONS: Vaccine Preventable Disease
Keywords: COVID-19; Vaccination
MeSH Terms: conditions — Vaccine-Preventable Diseases; COVID-19 | interventions — heterologous prime boost COVID-19 vaccination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: COVID-19 Vaccination — Receipt of full COVID-19 vaccination

SUMMARY:
This study will measure the levels of nasal mucosal Immunoglobulin A (IgA) and blood serum IgA up to one year after COVID vaccination, as well as examining what factors might affect antibody levels in the nose. This will be done through nasal epithelial lining fluid collection and standard venipuncture.

DETAILED DESCRIPTION:
Based on data demonstrating that SARS-CoV-2 infections results in virus-specific nasal IgA levels even in patients with mild infections and no/low serum antibody titers, we hypothesize that COVID vaccinations result in robust nasal IgA levels. Since previous data indicate that SARS-CoV2 specific IgA were transiently present following community-acquired infections, we will follow vaccine-induced nasal IgA levels over time (6-12 months). Our specific aims are as following:

Aim 1: Determine COVID vaccine specific immunoglobulin levels and immune mediator profiles in the nasal mucosa pre- and 14 days post second dose of COVID vaccine.

Aim 2: Determine COVID specific immunoglobulin levels and immune mediator profiles at 3, 6, and 12 months following complete vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Individuals at least 18 years of age who have or plan to receive a COVID-19 vaccination
* Able to be seen at UNC Chapel Hill's main campus up to 5 times in the next year

Exclusion Criteria:

* Individuals unwilling to give consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals vaccinated against COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Nasal Mucosal COVID-specific IgA | Up to 14 months
  Level of COVID-specific antibodies in the nasal mucosa
Serum COVID-specific IgA | Up to 14 months
  Level of COVID-specific antibodies in the blood serum

CONTACTS AND LOCATIONS:
Overall Officials: Ilona Jaspers, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No